CLINICAL TRIAL: NCT04412902
Title: Predictors of Recurrence for High Risk Endometrial Cancer Patients
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 109053-E
Record Dates: First submitted 2020-05-31; First posted 2020-06-02 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-04

CONDITIONS: High-risk Endometrial Cancer
MeSH Terms: interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: adjuvant therapy — Adjuvant chemotherapy and/or radiotherapy

SUMMARY:
This study will analyze whether there is any difference in recurrence and survival rates among the patients who received different adjuvant therapies.

DETAILED DESCRIPTION:
The incidence of endometrial cancer is gradually increasing nowaday. The postoperative treatment of high-risk endometrial cancer is also inconsistent. Besides, the recurrence of high-risk endometrial cancer is high.The investigators retrospective study will analyze the factors associated with recurrence of endometrial cancer, especially for different adjuvant therapies.

ELIGIBILITY:
Inclusion Criteria:

* All patients with high risk stage I endometrial cancer and all patients with stage II and stage III endometrial cancer and who underwent therapy in Far Eastern Memorial Hospital from 2009/01/01~2019/09/17.

Exclusion Criteria:

* Patients with stage I endometrial cancer do not have high risk factors.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — high risk endometrial cancer patients
Study Population: All high risk endometrial cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Factors affecting overall survival | 10 years
  Factors affecting overall survival

SECONDARY OUTCOMES:
Factors affecting progression-free survival | 10 years
  Factors affecting progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan